CLINICAL TRIAL: NCT04001348
Title: A Single-blind, Randomized, Uni-centre Study to Determine the Characteristics of Different Types of Safety Lancets on Blood Volume and Perceived Pain in Male and Female Volunteers
Brief Title: Characteristics of Different Types of Safety Lancets on Blood Volume and Perceived Pain in Male and Female Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mp05.13
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: safety lancets; lancet; capillary blood; capillary blood sampling; blood volume; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HTL-STREFA S.A.safety lancet type 610 (Experimental)
  Interventions: Device: Acti-Lance Lite; Device: Acti-Lance Universal; Device: Acti-Lance Special
- HTL-STREFA S.A.safety lancet type 553-556 (Experimental)
  Interventions: Device: Medlance Plus Super Lite; Device: Medlance Plus Lite; Device: Medlance Plus Universal; Device: Medlance Plus Extra; Device: Medlance Plus Special
- HTL-STREFA S.A.safety lancet type 430 (Experimental)
  Interventions: Device: Prolance Micro Flow; Device: Prolance Low Flow; Device: Prolance Normal Flow; Device: Prolance High Flow; Device: Prolance Max Flow; Device: Prolance Pediatric
- HTL-STREFA S.A.safety lancet type 520 (Experimental)
  Interventions: Device: MediSafe Solo 29 Gauge; Device: MediSafe Solo 23 Gauge

INTERVENTIONS:
Device: Acti-Lance Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Acti-Lance Universal — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Acti-Lance Special — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Medlance Plus Super Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 553-556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 553-556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Universal — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 553-556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Extra — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 553-556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Special — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 553-556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Prolance Micro Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Low Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Normal Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance High Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Max Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Pediatric — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: MediSafe Solo 29 Gauge — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 520
  Arms: HTL-STREFA S.A.safety lancet type 520
Device: MediSafe Solo 23 Gauge — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler. Perceived pain was assessed on the visual analog scale (VAS, numeric scale). VAS scale was assessed 5 minutes after the lancing procedure.
  Other Names: HTL-STREFA S.A.safety lancet type 520
  Arms: HTL-STREFA S.A.safety lancet type 520

SUMMARY:
The study was a randomized, single blind, uni-center pivotal study in male and female healthy volunteers, to determine capillary blood volume and pain perception obtained in a process of puncturing with different safety lancets.

A group of one hundred (100) healthy Caucasian male and female Subjects (aged > 18 to < 65 years old was randomized ) who were in good physical and mental condition. The Subjects had 4 (four) fingers (two fingers from each hand) lanced each with a different type of safety lancet. Overall, 4 (four) different safety lancets were investigated per each Subject.

Overall, 16 (sixteen) different safety lancets (4 different safety lancets per one Subject) were investigated, the capillary blood volume and pain were measured.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent.
* Male and female volunteers.
* Age between 18 and 65 inclusive.
* Able to communicate well with the Investigator and comply with the requirements of the study.
* Volunteers who are in good physical and mental health.

Exclusion Criteria:

* Pregnancy or breastfeeding (self-reported).
* Confirmed or suspected malignant cancer History of poor blood circulation.
* Any skin condition on his or her fingers that prevents blood sampling.
* Anxiety with needles or finger pricks.
* Clotting disorders (including bleeding) in medical history.
* Neuropathy or other condition affecting sensation in the hands.
* History of blood borne infection (e.g., HIV, hepatitis B or C, syphilis, malaria, babesiosis, brucellosis, leptospirosis, arboviral infections, relapsing fever, T lymphotropic virus Type 1, Creutzfeldt-Jakob disease).
* Currently participating in another study.
* History of drug or alcohol abuse within the 12 months prior to screening or evidence of such abuse.
* Intake of alcohol within 48 hours prior to the start of the study (self-reporting).
* Donation or loss of 400 mL or more of blood within 4 weeks prior to the start of the study.
* Any other condition that in the Investigator opinion may negatively influence Subject's participation in the study.
* Intake of medicines that affect blood coagulability (including anticoagulants such as vitamin K, antivirals and anticoagulants such as heparin, aspirin, thrombin inhibitors, vitamin K antagonists).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Volume (microliters) of blood in the capillary tube | The blood from the puncture site was collected to the capillaries by pressing during 2 minutes
  The amount of capillary blood volume collected after a single lancing of the fingertip.

SECONDARY OUTCOMES:
Pain perception: VAS | 5 minutes after lancing
  The intensity of pain perceived by the patient was assessed with the use of the numeric Visual Analog Scale (VAS). The Subject marked on the scale the number from 0 ("no pain") to 10 ("worst imaginable pain") that represented their perception of pain. A higher score indicated greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Monipol Clinical Pharmacology Research Centre, Krakow, Lesser Poland Voivodeship, Poland

REFERENCES:
- [Derived] Serafin A, Malinowski M, Prazmowska-Wilanowska A. Blood volume and pain perception during finger prick capillary blood sampling: are all safety lancets equal? Postgrad Med. 2020 Apr;132(3):288-295. doi: 10.1080/00325481.2020.1717160. Epub 2020 Feb 6. PMID 32027205